CLINICAL TRIAL: NCT04512144
Title: Mindfulness Practice in Endometrial and Cervical Cancers With Smartphone Applications (MECCA)
Brief Title: Mindfulness in Endometrial and Cervical Cancer
Acronym: MECCA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: St. Louis University (Other)
Responsible Party: Principal Investigator, Shannon Grabosch, MD, Assistant Professor of Gynecologic Oncology, St. Louis University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 30780
Record Dates: First submitted 2020-07-26; First posted 2020-08-13 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Gynecologic Cancer; Endometrial Cancer; Cervical Cancer; Quality of Life; Opioid Use
MeSH Terms: conditions — Endometrial Neoplasms; Uterine Cervical Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Patients with endometrial cancer will be approached for participation at their pre-operative visit. Patients with cervical cancer will be approached at their pre-treatment visit. If the patient opts to participate, she will be randomized to utilize the Headspace smartphone application or not. She will be provided a three month gift subscription. Headspace will be downloaded to her smartphone and she will be instructed on use. Patients will be asked to complete a quality of life survey on the day of enrollment, the day of surgery (endometrial cancer) or first brachytherapy (cervical cancer) and at their post-treatment visit. The patient will receive one phone call prior to her post-treatment visit requesting she bring her bottle of opiate pills with her for counting. The number of pills used will be recorded. The number of Headspace sessions will be recorded. An anonymous survey will be provided for completion. The patient will be provided a gift card at completion.
  Interventions: Behavioral: Headspace Smartphone Application
- Control (No Intervention): Patients with endometrial cancer will be approached for participation at their pre-operative visit. Patients with cervical cancer will be approached at their pre-treatment visit. If the patient opts to participate, she will be randomized to utilize the Headspace smartphone application or not. All patients in the control group may choose to practice calming or mindfulness exercises of their own accord but will not be specifically instructed to seek out such resources as is our standard practice. Patients will be asked to complete a quality of life survey on the day of enrollment, the day of surgery (endometrial cancer) or first brachytherapy (cervical cancer) and at their post-treatment visit. The patient will receive one phone call prior to her post-treatment visit requesting she bring her bottle of opiate pills with her for counting. The number of pills used will be recorded. An anonymous survey will be provided for completion. The patient will be provided a gift card at completion.

INTERVENTIONS:
Behavioral: Headspace Smartphone Application — Headspace is a smartphone application used for mindfulness, meditation, and stress reduction. It has been utilized in other behavioral and quality of life studies.
  Arms: Intervention

SUMMARY:
Patients with endometrial cancer who will be undergoing surgery or patients with cervical cancer who will be treated with chemoradiation will be randomized to utilize the Headspace smartphone application or not prior to their anticipated treatment.

DETAILED DESCRIPTION:
A diagnosis of cancer can be a major stress-inducing event. The prevalence of depression in patients diagnosed with cancer is estimated up to 16%. Practicing mindfulness is a cost-effective treatment which can also help manage treatment adverse effects and cancer-related symptoms.

Even short exposure and practice of mindfulness exercises have demonstrated improved subjective and objective measurements of stress and anxiety with breast biopsies. Patients with breast cancer also have improved quality of life with mindfulness training. Self-guided mindfulness with smartphone applications, specifically the app Headspace, has been associated with positive benefits and ease of use in the general population and among cancer patients.

A patient's inherent level of baseline mindfulness has been associated with lower pain scores following minimally invasive hysterectomy. This study did not specifically encourage practice of mindfulness exercises. Our own study of post-operative opiate usage in women following minimally invasive hysterectomy contains self-reported data of women using opiates to relax or help sleep. This suggests that mindfulness exercises may improve quality of life in these areas and thus reduce opiate usage. Patients undergoing minimally invasive hysterectomy for treatment of endometrial cancer were specifically chosen as a study cohort to build on our own data and that currently reported in the literature as well as the highest incidence of this cancer as a gynecologic malignancy. The second study cohort chosen was women with cervical cancer undergoing definitive treatment with chemo-sensitizing radiation given the significant endeavor required for complete treatment. Additionally, these women are often younger with the diagnosis of cervical cancer often being their first major medical diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* New diagnosis of either 1) endometrial cancer undergoing surgery or 2) cervical cancer undergoing chemo-sensitizing radiation
* Access to a smartphone

Exclusion Criteria:

* Non-English speaking
* No access to smartphone
* Current use of Headspace application

Ages: 18 Years to 90 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2020-07-25 (Actual); Primary Completion 2026-07-30 (Estimated); Study Completion 2026-07-30 (Estimated)

PRIMARY OUTCOMES:
Opiate Usage-Endometrial cancer | Enrollment to 30 days post op for endometrial cancer.
  The amount of opiates used during the acute (30 day) recovery after surgery for endometrial cancer or acute treatment with chemoradiation for cervical cancer will be recorded.
Opiate Usage-Cervical Cancer | Enrollment to 6 weeks post treatment for cervical cancer.
  The amount of opiates used during the acute treatment with chemoradiation for cervical cancer will be recorded.

SECONDARY OUTCOMES:
Five Facet Mindfulness Questionnaire | Enrollment to 4 weeks post op for endometrial cancer. Enrollment to 6 weeks post treatment for cervical cancer.
  Patients will be asked to complete a Five Facet Mindfulness Questionnaire form at enrollment, on the day of surgery (endometrial cancer) or first brachytherapy (cervical cancer), and at their post-treatment visit.
Functional Assessment of Cancer Therapy-General | Enrollment to 4 weeks post op for endometrial cancer. Enrollment to 6 weeks post treatment for cervical cancer.
  Patients will be asked to complete a Functional Assessment of Cancer Therapy-General form at enrollment, on the day of surgery (endometrial cancer) or first brachytherapy (cervical cancer), and at their post-treatment visit.
Complication Rates | Enrollment to 4 weeks post op for endometrial cancer. Enrollment to 6 weeks post treatment for cervical cancer.
  Surgical or treatment complications will be monitored in each group.
Patient satisfaction | Enrollment to 4 weeks post op for endometrial cancer. Enrollment to 6 weeks post treatment for cervical cancer.
  Patients from each group will be asked to complete an anonymous study-specific survey evaluating their satisfaction with the program.
Compliance | Enrollment to 4 weeks post op for endometrial cancer. Enrollment to 6 weeks post treatment for cervical cancer.
  The number of Headspace sessions utilized by patients in the intervention group will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Shannon Grabosch, MD, Principal Investigator — St. Louis University
Locations (1):
- Saint Louis University, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No